CLINICAL TRIAL: NCT06886035
Title: Effectiveness of Curcuminoids in Controlling Postoperative Pain Following Total Laparoscopic Hysterectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, prof dr, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M07
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Care; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Our clinical ERAS (Enhanced Recovery After Surgery) protocols were implemented to control patients without any additional intervention
- Study Group (Experimental): Our clinical ERAS (Enhanced Recovery After Surgery) protocols were implemented to study patients. The study group also began a regimen of 100 mg oral liposomal curcumin (administered as 50 mg twice daily) one day before the procedure. Following surgery, oral liposomal curcumin (50 mg twice daily) was restarted 8 hours postoperatively and maintained for an additional two days.
  Interventions: Drug: liposomal curcumin

INTERVENTIONS:
Drug: liposomal curcumin — The study group began a regimen of 100 mg oral liposomal curcumin (administered as 50 mg twice daily) one day prior to the procedure. Following surgery, oral liposomal curcumin (50 mg twice daily) was restarted 8 hours postoperatively and maintained for an additional two days. ( A total dose 300 mg)
  Arms: Study Group

SUMMARY:
Total hysterectomy is one of the most common surgical procedures in gynecology. Total laparoscopic hysterectomy (TLH) has several advantages over open surgery, such as better cosmetic outcomes, faster recovery, and an earlier return to normal activities and work, and has thus become the preferred approach Nonetheless, postoperative pain (PP) remains an issue of concern.

The reported incidence of PP after TLH ranges from 35 % to 63 %. The origin of PP after laparoscopy is multifactorial, arising from several perioperative factors, including pneumoperitoneum, stretching of the intraabdominal cavity, blood left in the abdomen, and dissection of the pelvic region. A prospective trial found more intense pain and greater analgesia requirement in the immediate postoperative period associated with laparoscopic surgery than with laparotomy. Methods to decrease the severity of PP are required before TLH can be confidently recommended.

Curcumin has several benefits, which are endorsed by the World Health Organization (WHO).

That is, it can be used to treat dyspepsia and peptic ulcer. Moreover, it has anti-inflammatory and analgesic properties. Most benefits are attributed to its anti-oxidant and anti-inflammatory effects. Curcuminoid is the active ingredient of turmeric. Curcuminoids are used in laparoscopic surgery because of their aforementioned benefits. Further, the use of traditional medicine, which is low-cost and effective in improving postoperative pain due to abdominal diştention, is assessed.

ELIGIBILITY:
Inclusion Criteria:

-Laparoscopic total hysterectomy and salpingectomy, with the option of additional procedures such as oophorectomy, uterosacral ligament plications, trans obturator tape insertion, or sentinel lymphadenectomy candidates

* They should be able to understand and sign an informed consent
* They should be literate enough to understand the maintenance of a diary recording pain scores, QoL-15 scores, and any adverse event

Exclusion Criteria:

* Patients with any peripheral or central neuropathic pain

  * Patients used to taking over-the-counter painkiller pills
  * Patients with a history of alcohol intake/drug dependence
  * Patients with a history of psychosis

    *Patients with chronic inflammatory diseases who cannot be taken off nonsteroidal anti-inflammatory drugs (NSAIDs)/painkillers
  * Patients on immunosuppressive/cytotoxic/steroid therapy. *Patients with a known allergy to duloxetine

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
the visual analogue scale (VAS) | 24 hours after surgery
  The primary goal was to assess the variation in postoperative pain levels recorded on the VAS (scored from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable) 24 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ariyasriwatana C, Phoolcharoen N, Oranratanaphan S, Worasethsin P. Efficacy of Curcuminoids in Managing Postoperative Pain after Total Laparoscopic Hysterectomy: A Randomized Controlled, Open-Label Trial. Complement Med Res. 2022;29(3):223-227. doi: 10.1159/000521669. Epub 2022 Jan 5. PMID 34986477
- [Background] Nurullahoglu KE, Okudan N, Belviranli M, Oz M. The comparison of preemptive analgesic effects of curcumin and diclofenac. Bratisl Lek Listy. 2014;115(12):757-60. doi: 10.4149/bll_2014_146. PMID 25520223